CLINICAL TRIAL: NCT02014467
Title: A Twelve-Month Randomized, Double-Blind, Placebo Controlled, Parallel-Group, Multicenter Study to Evaluate the Efficacy and Safety of Denosumab in Chinese Postmenopausal Women With Osteoporosis at Increased Risk of Fracture
Brief Title: Denosumab China Phase III Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 114165
Record Dates: First submitted 2013-12-12; First posted 2013-12-18 (Estimated); Results first posted 2016-10-31 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-09

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Denosumab; Calcium; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Denosumab 60mg (Experimental): injection
  Interventions: Drug: Denosumab; Dietary Supplement: Elemental Calcium; Dietary Supplement: Vitamin D
- Placebo (Placebo Comparator): injection
  Interventions: Drug: Placebo; Dietary Supplement: Elemental Calcium; Dietary Supplement: Vitamin D

INTERVENTIONS:
Drug: Denosumab — Injection
  Arms: Denosumab 60mg
Drug: Placebo — Injection
  Arms: Placebo
Dietary Supplement: Elemental Calcium — Oral, at least 600 mg
Dietary Supplement: Vitamin D — Oral, at least 400 IU

SUMMARY:
This study is to evaluate the efficacy and safety of denosumab 60 milligrams (mg) for 12 month treatment in Chinese postmenopausal women with osteoporosis at increased risk of fracture.

DETAILED DESCRIPTION:
The aim of this Phase III, randomized, double-blind, placebo-controlled, parallel-group study is to evaluate the efficacy and safety of denosumab (DMAb) in Chinese postmenopausal women with osteoporosis at increased risk of fracture. The study design consists of two phases: Screening and 12-month Double-Blind treatment phase. Following the Screening phase, all eligible subjects will be randomized to receive Double-Blind DMAb (60 mg) or Placebo study medication in a 3:1 ratio. DMAb 60 mg and placebo will be administered as a single subcutaneous (SC) injection at the beginning of the Double-Blind phase and at 6 months following the initial dose. All subjects will receive daily supplementation of oral elemental calcium (at least 600 mg) and vitamin D (at least 400 International Units [IU]). The primary objective is to determine the effects of DMAb compared to placebo with respect to mean percent change in BMD at the lumbar spine, as measured by dual-energy x-ray absorptiometry (DXA), from Baseline to Month 12. Secondary objectives include the evaluation between the DMAb and placebo treatment groups: change in BMD: at the lumbar spine (Month 6), total hip (Months 6 and 12), femoral neck (Months 6 and 12) and trochanter (Months 6 and 12); and serum biomarkers of bone formation and resorption (Months 6 and 12). Clinical safety of denosumab will also be assessed in this population.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing and able to provide written informed consent.
* Of Chinese origin - defined as being born in China, having four ethnic Chinese grandparents.
* Ambulatory woman between the age of 60 and 90 years, inclusive.
* The subject has a BMD absolute value consistent with a T-score<-2.5 and >-4.0 at either the lumbar spine or total hip.
* All subjects must have at least one of following additional the risk factors:

history of fracture parental history of hip fracture increased bone turnover rate at screening (s-CTX >1.0 SD above the mean in healthy premenopausal women) low body weight (BMI≤19kg/m2) elderly (age≥70y) current smoker

* Postmenopausal defined as >5 years postmenopausal, which can be >5 years of spontaneous amenorrhea or >5 years post surgical bilateral oophorectomy. Use follicle stimulating hormone (FSH) levels >40 mIU/mL to confirm surgical postmenopausal status, where bilateral oophorectomy status is uncertain.

Exclusion Criteria:

* Bone/metabolic disease:

Any metabolic bone disease, e.g., osteomalacia or osteogenesis imperfecta, which may interfere with the interpretation of the findings.

Paget's disease Cushing's disease Hyperprolactinemia

* Current hyperparathyroidism or hypoparathyroidism by medical record
* Thyroid condition: Hyperthyroidism or hypothyroidism. Only subjects with hypothyroidism who are on stable thyroid hormone replacement therapy may be allowed per the following criteria:

If TSH level is below normal range, subject is not eligible for the study. If TSH level is elevated (>5.5 μIU/mL and ≤10.0 μIU/mL), serum T4 should be measured.

If serum T4 is within normal range, subject is eligible. If serum T4 is outside of normal range, subject is not eligible for the study. If TSH level is > 10.0 μIU/mL, subject is not eligible.

* Rheumatoid arthritis
* Malignancy:

Malignancy (except fully resected cutaneous basal cell or squamous cell carcinoma, cervical or breast ductal carcinoma in situ) within the last 5years.

* Malabsorption syndrome: malabsorption syndrome or any gastrointestinal disorders associated with malabsorption, for example Crohn's Disease and chronic pancreatitis.
* Renal disease - severe renal impairment
* Liver disease:

Cirrhosis of the liver Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice), known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones). Chronic stable hepatitis B and C are acceptable if the subject otherwise meets study entry criteria (e.g., presence of hepatitis B surface antigen or positive Hepatitis C test result within 3 months of Screening).

* Drug or alcohol abuse: Evidence of alcohol or substance-abuse within the last 12 months which the investigator believes would interfere with understanding or completing the study.
* Biological abnormalities:

Any disorder that compromises the ability of the subject to give written informed consent or to comply with study procedures.

Any physical or psychiatric disorder which, in the opinion of the investigator, will prevent the subject from completing the study or interfere with the interpretation of the study results.

Known to have tested positive for human immunodeficiency virus (HIV).

* Vitamin D deficiency: Vitamin D deficiency (25-(OH) vitamin D level <20 ng/mL). Vitamin D repletion will be permitted and after repletion subjects may be re-tested once for 25-(OH) vitamin D levels.
* Oral/Dental Conditions Prior history or current evidence of osteomyelitis or osteonecrosis of the jaw. Active dental or jaw condition which requires oral surgery. Planned invasive dental procedure. Non-healed dental or oral surgery.

Concomitant Medications:

* Previous strontium or IV bisphosphonate: Administration of intravenous (IV) bisphosphonate, fluoride, or strontium for osteoporosis within the last 5 years.
* Oral bisphosphonate: Oral bisphosphonate treatment for osteoporosis:

If used for ≥3 years cumulatively, subject is ineligible.

If used for >3-months but <3 years cumulatively:

If the last dose was <1 year before enrolment, subject is ineligible. If the last dose was ≥1 year before enrolment, subject is eligible. If used ≤3 months, cumulatively, subject is eligible.

* Bone metabolism drugs: Administration of any of the following treatments within the last 6 weeks:

Parathyroid hormone (PTH) or PTH derivatives, e.g., teriparatide. Anabolic steroids or testosterone. Glucocorticosteroids (>5 mg prednisone equivalent per day for more than 10 days).

Systemic hormone replacement therapy. Selective estrogen receptor modulators (SERMs), e.g., raloxifene Tibolone. Calcitonin. Calcitriol or vitamin D derivatives. Other bone active drugs including anti-convulsives (except benzodiazepines) and heparin.

Chronic systemic ketoconazole, androgens, ACTH, cinacalcet, aluminum, lithium, protease inhibitors, methotrexate, gonadotropin-releasing hormone agonists.

* Investigational drug exposure: Currently enrolled in an investigational device or drug trial(s) or it has not been at least 30 days since the last study visit in an investigational device or drug trial(s), or subject is receiving other investigational agent(s).
* Sensitivity: Known sensitivity to mammalian cell-derived drug products.
* Clinically significant hypersensitivity to denosumab Abnormal laboratory values
* General: Any laboratory abnormality which, in the opinion of the investigator, will prevent the subject from completing the study or interfere with the interpretation of the study results.
* Abnormal serum calcium: current hypocalcemia or hypercalcemia. Albumin adjusted serum calcium levels must be within normal limits of the central laboratory.
* Liver transaminases:

Serum aspartate aminotransferase (AST) ≥2.0 x upper limits of normal (ULN). Serum alanine aminotransferase (ALT) ≥2.0 x ULN. Alkaline phosphatase and bilirubin ≥1.5 x ULN (isolated bilirubin ≥1.5 ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%.

* DXA measurements:

Less than two lumbar vertebrae evaluable for DXA measurements. Height, weight, or girth which may preclude accurate DXA measurements.

* Subjects with a history of greater than 2 vertebral fractures.
* Subjects at very high risk of fracture who must be treated with active drugs in the opinion of investigator.

Ages: 60 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 486 (Actual)
Dates: Start 2014-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- China (4):
  - GSK Investigational Site, Chengdu, Sichuan
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Chengdu
  - GSK Investigational Site, Shanghai

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study design consists of two phases: Screening Phase and 12-month Double-blind Treatment Phase. The Screening Phase was to last up to a maximum of 2.5 months, which was followed by a 12-month Double-blind Treatment Phase. The total participation time in the study was approximately 14.5 months.
Pre-assignment Details: A total of 909 participants were screened, of whom 485 were randomized in a 3: 1 ratio to receive one of the two study treatments. A total of 484 participants received at least single dose of investigational product (IP).
Groups:
- Denosumab 60 mg: Participants received single subcutaneous (SC) injection of denosumab 60 milligrams (mg) at Baseline and Month 6 during the Double-blind Treatment Phase. Particpants also received daily oral supplementation of elemental calcium (at least 600 mg) and vitamin D (at least 400 international unit [IU]).
- Placebo: Participants received single SC injection of placebo at Baseline and Month 6 during the Double-blind Treatment Phase.Participants also received daily oral supplementation of elemental calcium (at least 600 mg) and vitamin D (at least 400 IU).
Period: Overall Study
Arm/Group | Denosumab 60 mg | Placebo
Started | 365 | 119
Completed | 340 | 112
Not Completed | 25 | 7
Not completed — Adverse Event | 4 | 0
Not completed — Protocol Violation | 3 | 0
Not completed — Physician Decision | 2 | 3
Not completed — Withdrawal by Subject | 16 | 4

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received single SC injection of placebo at Baseline and Month 6 during the Double-blind Treatment Phase. Participants also received daily oral supplementation of elemental calcium (at least 600 mg) and vitamin D (at least 400 IU).
- Total: Total of all reporting groups
Arm/Group | Denosumab 60 mg | Placebo | Total
Number analyzed (Participants) | 365 | 119 | 484
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.9 (6.10) | 69.6 (5.75) | 69.0 (6.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 365 | 119 | 484
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - East Asian Heritage | 365 | 119 | 484

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Bone Mineral Density (BMD) at the Lumbar Spine at Month 12
Description: Bone mineral density (BMD) is the amount of bone mineral in bone tissue. BMD scan was done using dual energy x-ray absorptiometry (DXA). It is used to identify osteoporosis, determine risk for fractures, and measure response to osteoporosis treatment. The percentage change from Baseline for BMD was calcuated as the value at the indicated time point minus the Baseline value multiplied by 100 and divided by the Baseline value. The analysis was performed by Analysis of Covariance (ANCOVA) model adjusted for treatment, region and Baseline BMD for the skeletal site under consideration as a continuous covariate for assessment. Region and treatment by region interaction was included in the model. Screening visit was considered as Baseline for BMD. For participants who withdrew early, the missing BMD assessments was estimated by the Last Observation Carried Forward (LOCF), provided the assessment was taken on or after at least one month on-therapy.
Time Frame: Baseline and Month 12
Population: Intent-to-Treat (ITT) Population: all safety Population participants (consisting of all participants who received at least one dose of study medication) who had a Baseline and at least one valid post-Baseline efficacy measure. Participants with values at Baseline and Month 12 were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 350 | 116
Percentage change | 5.22 (0.274) | 0.79 (0.391)
Statistical Analysis 1: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = 4.42, 95% CI 2-sided [3.67 to 5.18]
Statistical Analysis 2: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p = 0.7495, ANCOVA — Treatment By Region Interaction: Based on ANCOVA, Percent change from Baseline = Baseline + treatment + region + treatment by region

2. Secondary Outcome: Percent Change From Baseline in BMD at the Lumbar Spine at Month 6
Description: BMD is the amount of bone mineral in bone tissue. BMD scan was done using DXA. It is used to identify osteoporosis, determine risk for fractures, and measure response to osteoporosis treatment. The percentage change from Baseline for BMD was calculated as the value at the indicated time point minus the Baseline value multiplied by 100 and divided by the Baseline value. ANCOVA model adjusted for treatment, center/region and Baseline BMD for the skeletal site under consideration as a continuous covariate for assessment. Region and treatment by region interaction was included in the model. Screening visit was considered as baseline for BMD. For participants who withdrew early, the missing BMD assessments was estimated by the LOCF, provided the assessment was taken on or after at least one month on-therapy.
Time Frame: Baseline and Month 6
Population: ITT Population. Participants with values at Baseline and Month 6 were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 350 | 116
Percentage change | 3.77 (0.273) | 0.57 (0.390)
Statistical Analysis 1: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = 3.21, 95% CI 2-sided [2.45 to 3.96]
Statistical Analysis 2: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p = 0.9029, ANCOVA — [p-value comment as in outcome 1, analysis 2]

3. Secondary Outcome: Percent Change From Baseline in BMD at the Total Hip at Month 6
Description: as for outcome 2
Time Frame: Baseline and Month 6
Population: ITT Population. Participants with values at Baseline and Month 6 were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 347 | 115
Percentage change | 2.36 (0.193) | 0.11 (0.279)
Statistical Analysis 1: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = 2.26, 95% CI 2-sided [1.72 to 2.80]
Statistical Analysis 2: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p = 0.1070, ANCOVA — [p-value comment as in outcome 1, analysis 2]

4. Secondary Outcome: Percent Change From Baseline in BMD at the Femoral Neck at Month 6
Description: as for outcome 2
Time Frame: Baseline and Month 6
Population: ITT Population. Participants with values at Baseline and Month 6 were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 347 | 115
Percentage change | 1.91 (0.219) | 0.32 (0.315)
Statistical Analysis 1: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = 1.59, 95% CI 2-sided [0.98 to 2.20]
Statistical Analysis 2: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p = 0.4369, ANCOVA — [p-value comment as in outcome 1, analysis 2]

5. Secondary Outcome: Percent Change From Baseline in BMD at the Trochanter at Month 6
Description: as for outcome 2
Time Frame: Baseline and Month 6
Population: ITT Population. Participants with values at Baseline and Month 6 were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 347 | 115
Percentage change | 2.76 (0.344) | -0.59 (0.498)
Statistical Analysis 1: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = 3.36, 95% CI [2.39 to 4.32]
Statistical Analysis 2: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p = 0.6082, ANCOVA — [p-value comment as in outcome 1, analysis 2]

6. Secondary Outcome: Percent Change From Baseline in BMD at the Total Hip at Month 12
Description: as for outcome 2
Time Frame: Baseline and Month 12
Population: ITT Population. Participants with values at Baseline and Month 12 were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 348 | 115
Percentage change | 3.03 (0.202) | -0.28 (0.293)
Statistical Analysis 1: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = 3.31, 95% CI 2-sided [2.74 to 3.88]
Statistical Analysis 2: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p = 0.3513, ANCOVA — [p-value comment as in outcome 1, analysis 2]

7. Secondary Outcome: Percent Change From Baseline in BMD at the Femoral Neck at Month 12
Description: as for outcome 2
Time Frame: Baseline and Month 12
Population: ITT Population. Participants with values at Baseline and Month 12 were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 348 | 115
Percentage change | 2.77 (0.233) | 0.16 (0.337)
Statistical Analysis 1: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = 2.62, 95% CI 2-sided [1.96 to 3.27]
Statistical Analysis 2: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p = 0.5410, ANCOVA — [p-value comment as in outcome 1, analysis 2]

8. Secondary Outcome: Percent Change From Baseline in BMD at the Trochanter at Month 12
Description: as for outcome 2
Time Frame: Baseline and Month 12
Population: ITT Population. Participants with values at Baseline and Month 12 were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 348 | 115
Percentage change | 3.88 (0.356) | -0.83 (0.517)
Statistical Analysis 1: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = 4.72, 95% CI 2-sided [3.71 to 5.72]
Statistical Analysis 2: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p = 0.3957, ANCOVA — [p-value comment as in outcome 1, analysis 2]

9. Secondary Outcome: Percent Change in Serum Carboxy-terminal Cross-linking Telopeptide of Type I Collagen (s-CTX) From Baseline to Month 6 and Month 12
Description: s-CTX is biomarker of bone resorption and formation. s-CTX was assessed during Screening, Month 6 and Month 12 in the Double-blind Treatment Phase. The value during Screening was considered as the Baseline value. Percent change from Baseline was assessed as the value at the indicated visit minus the Baseline value divided by the Baseline value x 100. A two-sided Wilcoxon rank sum test was used to compare percent change in s-CTX. Between group inferences is presented by p-values, Hodges-Lehmann estimates along with 95% confidence intervals.
Time Frame: Baseline, Month 6 and Month 12
Population: ITT Population. Only those participants with values at Baseline and Month 6 and Month 12 are included in the analysis (represented by n=X, X in the category titles).
Measure: Median (Inter-Quartile Range); unit: Percentage change
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 354 | 117
Percentage change
  s-CTX, Month 6, n=353, 117 | -79.20 [-86.80 to -66.45] | -19.35 [-35.97 to -2.74]
  s-CTX, Month 12, n=335, 108 | -64.51 [-77.29 to -38.52] | -5.94 [-29.52 to 16.67]
Statistical Analysis 1: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum test — Two-Sided, Wilcoxon t Approximation; Hodges Lehmann Estimate of Difference = -56.92, 95% CI 2-sided [-61.38 to -52.65] — s-CTX at Month 6
Statistical Analysis 2: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum test — Two-Sided, Wilcoxon t Approximation; Hodges Lehmann Estimate of Difference = -52.56, 95% CI [-59.38 to -46.17] — s-CTX at Month 12

10. Secondary Outcome: Percent Change in Serum Procollagen Type I N Propeptideserum (s-PINP) From Baseline to Month 6 and Month 12
Description: s-PINP is biomarker of bone resorption and formation. s-PINP was assessed during Screening, Month 6 and Month 12 in the Double-blind Treatment Phase. The value during Screening was considered as the Baseline value. Percent change from Baseline was assessed as the value at the indicated visit minus the Baseline value divided by the Baseline value x 100. A two-sided Wilcoxon rank sum test was used to compare percent change in serum CTX. Between group inferences is presented by p-values, Hodges-Lehmann estimates along with 95% confidence intervals.
Time Frame: Baseline, Month 6, Month 12
Population: ITT Population: Only those participants with values at Baseline and Month 6 and Month 12 are included in the analysis (represented by n=X, X in the category titles).
Measure: Median (Inter-Quartile Range); unit: Percentage change
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 352 | 117
Percentage change
  s-PINP, Month 6, n=352, 117 | -73.12 [-81.03 to -62.81] | -12.37 [-29.58 to 4.37]
  s-PINP, Month 12, n=335, 108 | -66.14 [-76.04 to -50.75] | -14.83 [-27.84 to 11.26]
Statistical Analysis 1: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum test — Two-Sided, Wilcoxon t Approximation; Hodges Lehmann Estimate of Difference = -56.94, 95% CI 2-sided [-61.60 to -52.70] — s-PINP at Month 6
Statistical Analysis 2: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum test — Two-Sided, Wilcoxon t Approximation; Hodges Lehmann Estimate of Difference = -51.21, 95% CI 2-sided [-56.26 to -45.91] — s-PINP at Month 12

11. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at Month 1, Month 3, Month 6, and Month 12
Description: Baseline value was obtained at Randomization (Visit 3). If missing, the most recent non-missing value was used. Change in Baseline value was assessed as the value at the indicated visit minus the Baseline value. Change from Baseline in SBP and DBP was assessed at Baseline, Month 1, Month 3, Month 6, and Month 12.
Time Frame: Baseline, Month 1, Month 3, Month 6 and Month 12
Population: Safety Population: all participants who received at least one dose of study medication. Two participants randomized to placebo group received denosumab by mistake. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 367 | 117
Millimeters of mercury (mmHg)
  SBP, Month 1, n = 365, 117 | -1.8 (11.01) | -1.3 (11.89)
  SBP, Month 3, n = 362, 117 | -3.4 (12.62) | -0.5 (12.16)
  SBP, Month 6, n = 350, 114 | 0.1 (12.76) | 1.5 (13.25)
  SBP, Month 12, n = 342, 110 | -0.5 (11.83) | -0.1 (11.69)
  DBP, Month 1, n = 365, 117 | 0.0 (6.95) | 0.6 (7.58)
  DBP, Month 3, n = 362, 117 | -1.5 (7.70) | 0.2 (6.50)
  DBP, Month 6, n = 350, 114 | -0.3 (7.67) | 1.1 (8.34)
  DBP, Month 12, n = 342, 110 | 0.2 (7.63) | 1.2 (7.75)

12. Secondary Outcome: Change From Baseline in Heart Rate at Month 1, Month 3, Month 6, and Month 12
Description: Baseline value was obtained at Randomization (Visit 3). If missing, the most recent non-missing value was used. Change in Baseline value was assessed as the value at the indicated visit minus the Baseline value. Change from Baseline in heart rate was assessed at Baseline, Month 1, Month 3, Month 6 and Month 12.
Time Frame: Baseline, Month 1, Month 3, Month 6 and Month 12
Population: Safety Population. Two participants randomized to placebo group received denosumab by mistake. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 367 | 117
Beats per minute
  Heart Rate, Month 1, n = 365, 117 | -0.8 (6.88) | -2.1 (7.51)
  Heart Rate, Month 3, n = 362, 117 | 1.2 (10.28) | 0.2 (9.08)
  Heart Rate, Month 6, n = 350, 114 | -0.4 (8.23) | -1.3 (9.01)
  Heart Rate, Month 12, n = 342, 110 | -0.9 (7.55) | 0.1 (10.48)

13. Secondary Outcome: Change From Baseline in Alanine Amino Transferase, Alkaline Phosphatase, Aspartate Amino Transferase, and Gamma Glutamyl Transferase at Month 1, Month 6 and Month 12
Description: Baseline values were obtained at Screening (Visit 2). If missing, the most recent non-missing value was used. Change in Baseline value was assessed as the value at the indicated visit minus the Baseline value. Blood samples were collected for measurement. Alanine amino transferase, alkaline phosphatase, aspartate amino transferase, and gamma glutamyl transferase were assessed at Baseline, Month 1, Month 6 and Month 12.
Time Frame: Baseline, Month 1, Month 6, and Month 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: International unit per liter (IU/L)
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 367 | 117
International unit per liter (IU/L)
  Alanine Amino Transferase, Month 1, n = 365, 117 | 0.2 (6.27) | -0.1 (5.91)
  Alanine Amino Transferase, Month 6, n = 350, 114 | 1.9 (9.00) | 0.7 (7.19)
  Alanine Amino Transferase, Month 12, n = 340, 109 | 1.5 (12.49) | 0.2 (8.45)
  Alkaline Phosphatase, Month 1, n = 365, 117 | -3.3 (11.00) | -3.2 (10.03)
  Alkaline Phosphatase, Month 6, n = 350, 114 | -21.0 (17.20) | -1.2 (11.43)
  Alkaline Phosphatase, Month 12, n = 340, 109 | -23.4 (17.36) | -5.3 (11.06)
  Aspartate Amino Transferase, Month 1, n = 365, 117 | -0.1 (4.34) | -0.4 (4.41)
  Aspartate Amino Transferase, Month 6, n = 350, 114 | 1.2 (7.84) | 0.2 (5.28)
  Aspartate Amino Transferase,Month 12, n = 340, 109 | 0.1 (7.41) | -0.8 (5.94)
  Gamma Glutamyl Transferase, Month 1, n = 365, 117 | 0.2 (11.52) | -0.6 (5.82)
  Gamma Glutamyl Transferase, Month 6, n = 350, 114 | 0.1 (11.22) | -0.1 (6.44)
  Gamma Glutamyl Transferase, Month 12, n = 340, 109 | -0.9 (9.96) | 0.3 (10.09)

14. Secondary Outcome: Change From Baseline in Creatine Kinase, Lactate Dehydrogenase at Month 6 and Month 12.
Description: Baseline values was obtained at Screening (Visit 2). If missing, the most recent non-missing value was used. Change in Baseline value was assessed as the value at the indicated visit minus the Baseline value. Blood samples were collected for measurement. Creatine kinase and lactate dehydrogenase were assessed at Baseline, Month 6 and Month 12.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: International unit per liter (IU/L)
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 367 | 117
International unit per liter (IU/L)
  Creatine Kinase, Month 6, n = 350, 114 | -3.7 (43.41) | -3.7 (31.64)
  Creatine Kinase, Month 12, n = 340, 109 | -2.6 (53.83) | -0.3 (38.58)
  Lactate Dehydrogenase, Month 6, n = 350, 114 | -3.4 (19.62) | -5.6 (19.60)
  Lactate Dehydrogenase, Month 12, n = 340, 109 | -2.2 (18.50) | -4.0 (23.16)

15. Secondary Outcome: Change From Baseline in Albumin at Month 1, Month 6 and Month 12.
Description: Baseline value was obtained at Screening (Visit 2). If missing, the most recent non-missing value was used. Change in Baseline value was assessed as the value at the indicated visit minus the Baseline value. Blood samples were collected for measurement. Albumin was assessed at Baseline, Month 1, Month 6 and Month 12.
Time Frame: Baseline, Month 1, Month 6 and Month 12.
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Gram per liter (G/L)
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 367 | 117
Gram per liter (G/L)
  Albumin, Month 1, n = 365, 117 | -0.6 (1.93) | -0.7 (1.75)
  Albumin, Month 6, n = 350, 114 | 0.7 (1.96) | 0.5 (2.09)
  Albumin, Month 12, n = 340, 109 | 0.2 (1.82) | 0.1 (2.11)

16. Secondary Outcome: Change From Baseline in Globulin at Month 6 and Month 12.
Description: Baseline value was obtained at Screening (Visit 2). If missing, the most recent non-missing value was used. Change in Baseline value was assessed as the value at indicated visit minus the Baseline value. Blood samples were collected for measurement. Globulin was assessed at Baseline, Month 6 and Month 12.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Grams per liter (G/L)
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 367 | 117
Grams per liter (G/L)
  Globulin, Month 6, n = 350, 114 | -0.3 (2.29) | -0.2 (2.35)
  Globulin, Month 12, n = 340, 109 | -0.5 (2.57) | -0.4 (2.78)

17. Secondary Outcome: Change From Baseline in Hemoglobin and Total Protein at Month 6 and Month 12.
Description: Baseline value was obtained at Screening (Visit 2). If missing, the most recent non-missing value was used. Change in Baseline value was assessed as the value at indicated visit minus the Baseline value. Blood samples were collected for measurement. Hemoglobin and total protein were assessed at Baseline, Month 6 and Month 12.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Grams per liter (G/L)
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 367 | 117
Grams per liter (G/L)
  Hemoglobin, Month 6, n = 346, 113 | 2.3 (5.33) | 1.9 (5.54)
  Hemoglobin, Month 12, n = 339, 109 | 0.2 (6.12) | 0.7 (6.52)
  Total Protein, Month 6, n = 350, 114 | 0.4 (3.30) | 0.3 (3.34)
  Total Protein, Month 12, n = 340, 109 | -0.2 (3.57) | -0.3 (3.60)

18. Secondary Outcome: Change From Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes, Platelet Count, Total Neutrophils-total Absolute Neutrophil Count (ANC), White Blood Cell Count at Month 6 and Month 12.
Description: Baseline value was obtained at Screening (Visit 2). If missing, the most recent non-missing value was used. Change in Baseline value was assessed as the value at the indicated visit minus the Baseline value. Blood samples were collected for measurement. Basophils, eosinophils, lymphocytes, monocytes, platelet count, total neutrophils-total ANC and white blood cell count were assessed at Baseline, Month 6 and Month 12.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Giga per liter (GI/L)
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 367 | 117
Giga per liter (GI/L)
  Basophils, Month 6, n = 346, 113 | -0.002 (0.0180) | -0.001 (0.0180)
  Basophils, Month 12, n = 339, 109 | -0.001 (0.0160) | -0.003 (0.0183)
  Eosinophils, Month 6, n = 346, 113 | 0.025 (0.1402) | 0.013 (0.1240)
  Eosinophils, Month 12, n = 339, 109 | -0.001 (0.1530) | 0.006 (0.1382)
  Lymphocytes, Month 6, n = 346, 113 | 0.011 (0.3658) | -0.020 (0.3513)
  Lymphocytes, Month 12, n = 339, 109 | -0.064 (0.3689) | -0.082 (0.3584)
  Monocytes, Month 6, n = 346, 113 | 0.042 (0.0999) | 0.035 (0.0868)
  Monocytes, Month 12, n = 339, 109 | -0.007 (0.1002) | -0.004 (0.0800)
  Platelet count, Month 6, n = 345, 113 | 3.0 (30.49) | -0.1 (24.08)
  Platelet count, Month 12, n = 337, 109 | -6.8 (26.66) | -3.6 (30.82)
  Total ANC, Month 6, n = 346, 113 | 0.153 (1.0436) | -0.002 (0.8814)
  Total ANC, Month 12, n = 339, 109 | -0.071 (0.9412) | -0.119 (0.9691)
  White Blood Cell count, Month 6, n = 346, 113 | 0.23 (1.166) | 0.02 (1.036)
  White Blood Cell count, Month 12, n = 339, 109 | -0.14 (1.083) | -0.20 (1.164)

19. Secondary Outcome: Change From Baseline in Calcium (Corrected), Calcium at Month 1, Month 6 and Month 12.
Description: Baseline value was obtained at Screening (Visit 2). If missing, the most recent non-missing value was used. Change in Baseline value was assessed as the value at the indicated visit minus the Baseline value. Blood samples were collected for measurement. Calcium (corrected) and calcium were assessed at Baseline, Month 1, Month 6 and Month 12.
Time Frame: Baseline, Month 1, Month 6 and Month 12.
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 367 | 117
Millimoles per liter (mmol/L)
  Calcium (corrected), Month 1, n = 365, 117 | -0.063 (0.0740) | 0.000 (0.0505)
  Calcium (corrected), Month 6, n = 350, 114 | -0.020 (0.0704) | -0.001 (0.0537)
  Calcium (corrected), Month 12, n = 340, 109 | -0.002 (0.0680) | -0.001 (0.0488)
  Calcium, Month 1, n = 365, 117 | -0.074 (0.0906) | -0.014 (0.0614)
  Calcium, Month 6, n = 350, 114 | -0.006 (0.0809) | 0.009 (0.0703)
  Calcium, Month 12, n = 340, 109 | 0.002 (0.0807) | 0.001 (0.0648)

20. Secondary Outcome: Change From Baseline in Chloride, Cholesterol, Glucose, Magnesium, Inorganic Phosphorous, Potassium, Sodium, Triglycerides, Urea/Blood Urea Nitrogen (BUN) at Month 6 and Month 12.
Description: Baseline value was obtained at Screening (Visit 2). If missing, the most recent non-missing value was used. Change in Baseline value was assessed as the value at the indicated visit minus the Baseline value. Blood samples were collected for measurement. Chloride, cholesterol, glucose, magnesium, inorganic phosphorous, potassium, sodium, triglycerides and urea/BUN were assessed at Baseline, Month 6 and Month 12.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 367 | 117
Millimoles per liter (mmol/L)
  Chloride, Month 6, n = 350, 114 | -0.9 (2.48) | -0.7 (2.37)
  Chloride, Month 12, n = 340, 109 | 0.4 (2.17) | 0.6 (2.34)
  Cholesterol, Month 6, n = 350, 114 | 0.039 (0.7626) | 0.057 (0.7837)
  Cholesterol, Month 12, n = 340, 109 | 0.047 (0.8909) | 0.058 (0.7889)
  Glucose, Month 6, n = 350, 114 | 0.12 (0.882) | 0.04 (1.052)
  Glucose, Month 12, n = 340, 109 | 0.16 (0.124) | -0.07 (0.752)
  Magnesium, Month 6, n = 350, 114 | 0.003 (0.0523) | -0.002 (0.0547)
  Magnesium, Month 12, n = 340, 109 | 0.013 (0.0485) | 0.012 (0.0572)
  Phosphorus, inorganic, Month 6, n = 350, 114 | -0.082 (0.1440) | -0.030 (0.1353)
  Phosphorus, inorganic, Month 12, n = 340, 109 | -0.063 (0.1520) | -0.028 (0.1304)
  Potassium, Month 6, n = 350, 114 | 0.00 (0.328) | 0.02 (0.294)
  Potassium, Month 12, n = 340, 109 | 0.01 (0.300) | -0.01 (0.294)
  Sodium, Month 6, n = 350, 114 | -0.8 (1.94) | -0.4 (2.24)
  Sodium, Month 12, n = 340, 109 | -1.3 (1.93) | -0.7 (1.76)
  Triglycerides, Month 6, n = 350, 114 | -0.082 (0.7604) | -0.000 (0.6753)
  Triglycerides, Month 12, n = 340, 109 | -0.014 (0.9367) | -0.029 (0.7489)
  Urea/BUN, Month 6, n = 350, 114 | -0.18 (1.045) | -0.35 (1.288)
  Urea/BUN, Month 12, n = 340, 109 | 0.04 (1.124) | 0.01 (1.466)

21. Secondary Outcome: Change From Baseline in Direct Bilirubin, Total Bilirubin at Month 1, Month 6 and Month 12.
Description: Baseline value was obtained at Screening (Visit 2). If missing, the most recent non-missing value was used. Change in Baseline value was assessed as the value at the indicated visit minus the Baseline value. Blood samples were collected for measurement. Direct bilirubin and total bilirubin were assessed at Baseline, Month 1, Month 6 and Month 12.
Time Frame: Baseline, Month 1, Month 6 and Month 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Micromoles per liter (UMOL/L)
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 367 | 117
Micromoles per liter (UMOL/L)
  Direct Bilirubin, Month 1, n = 365, 117 | -0.1 (0.67) | 0.1 (0.52)
  Direct Bilirubin, Month 6, n = 350, 114 | 0.0 (0.72) | 0.1 (0.66)
  Direct Bilirubin, Month 12, n = 340, 109 | 0.1 (0.67) | 0.2 (0.68)
  Total Bilirubin, Month 1, n = 365, 117 | -0.3 (2.83) | 0.2 (2.61)
  Total Bilirubin, Month 6, n = 350, 114 | 0.1 (2.91) | 0.2 (2.66)
  Total Bilirubin, Month 12, n = 340, 109 | 0.3 (2.98) | 0.2 (2.80)

22. Secondary Outcome: Change From Baseline in Creatinine and Uric Acid at Month 6 and Month 12
Description: Baseline value was obtained at Screening (Visit 2). If missing, the most recent non-missing value was used. Change in Baseline value was assessed as the value at the indicated visit minus the Baseline value. Blood samples were collected for measurement. Creatinine and uric acid were assessed at Baseline, Month 6 and Month 12.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Micromoles per liter (UMOL/L)
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 367 | 117
Micromoles per liter (UMOL/L)
  Creatinine, Month 6, n = 350, 114 | -0.47 (5.067) | -0.90 (5.611)
  Creatinine, Month 12, n = 340, 109 | -0.18 (5.116) | -0.30 (6.185)
  Uric acid, Month 6, n = 350, 114 | -8.9 (48.33) | -8.9 (48.58)
  Uric acid, Month 12, n = 340, 109 | -6.7 (49.84) | -2.7 (44.85)

23. Secondary Outcome: Change From Baseline in Hematocrit at Month 6 and Month 12.
Description: Baseline value was obtained at Screening (Visit 2). If missing, the most recent non-missing value was used. Change in Baseline value was assessed as the value at the indicated visit minus the Baseline value. Blood samples were collected for measurement. Hematocrit was assessed at Baseline, Month 6 and Month 12.
Time Frame: Baseline, Month 6 and Month 12.
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 367 | 117
Ratio
  Hematocrit, Month 6, n = 346, 113 | 0.0024 (0.01612) | 0.0012 (0.01662)
  Hematocrit, Month 12, n = 339, 109 | 0.0064 (0.01884) | 0.0079 (0.01926)

24. Secondary Outcome: Change From Baseline in Mean Corpuscle Hemoglobin at Month 6 and Month 12.
Description: Baseline value was obtained at Screening (Visit 2). If missing, the most recent non-missing value was used. Change in Baseline value was assessed as the value at the indicated visit minus the Baseline value. Blood samples were collected for measurement. Mean corpuscle hemoglobin was assessed at Baseline, Month 6 and Month 12.
Time Frame: Baseline, Month 6 and Month 12.
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Picograms (PG)
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 367 | 117
Picograms (PG)
  Mean Corpuscle Hemoglobin, Month 6, n = 346, 113 | 0.22 (0.599) | 0.18 (0.561)
  Mean Corpuscle Hemoglobin, Month 12, n = 339, 109 | -0.31 (0.691) | -0.38 (0.600)

25. Secondary Outcome: Change From Baseline in Mean Corpuscle Volume at Month 6 and Month 12.
Description: Baseline value was obtained at Screening (Visit 2). If missing, the most recent non-missing value was used. Change in baseline value was assessed as the value at the indicated visit minus the Baseline value. Blood samples were collected for measurement. Mean corpuscle volume was assessed at Baseline, Month 6 and Month 12.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Femtoliter (FL)
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 367 | 117
Femtoliter (FL)
  Mean Corpuscle Volume, Month 6, n = 346, 113 | -0.4 (1.77) | -0.5 (2.17)
  Mean Corpuscle Volume, Month 12, n = 339, 109 | 0.4 (2.01) | 0.3 (1.77)

26. Secondary Outcome: Change From Baseline in Red Blood Cell Count at Month 6 and Month 12
Description: Baseline value was obtained at screening (visit 2). If missing, the most recent non-missing value was used. Change in baseline value was assessed as: Value at Indicated visit minus Baseline value. Blood samples were collected for measurement. Red blood cell count was assessed at Baseline, Month 6 and Month 12.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Trillion cells per liter (TI/L)
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 367 | 117
Trillion cells per liter (TI/L)
  Red Blood Cell count, Month 6, n = 346, 113 | 0.04 (0.180) | 0.04 (0.170)
  Red Blood Cell count, Month 12, n = 339, 109 | 0.05 (0.203) | 0.07 (0.200)

27. Secondary Outcome: Number of Participants With Confirmed Anti-denosumab Antibody Formation at Baseline and Month 12
Description: Anti-denosumab antibody formation was assessed at Baseline (Visit 3) and Month 12. Binding antibody and neutralizing antibody assays were used to assess number of participants with anti-denosumab antibody.
Time Frame: Baseline and Month 12
Population: as for outcome 12
Measure: Number; unit: Participants
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 367 | 117
Participants
  Binding antibody detection, Baseline, n = 15, 3 | 0 | 0
  Binding antibody detection, Month 12, n = 29, 3 | 1 | 0
  Neutralising antibody detection,Month 12, n = 1,0 | 0 | 0

28. Secondary Outcome: Number of Participants With Any Adverse Events (AEs), Serious Adverse Events (Non-fatal Serious Adverse Events and Fatal Serious Adverse Events)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. A serious adverse event (SAE) is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or other events that may jeopardize the participant or may require medical or surgical intervention to prevent one of the outcome listed above, liver injury and impaired liver function and grade 4 laboratory abnormalities. Number of participants with any AEs, serious non-fatal AEs, serious fatal AEs have been presented.
Time Frame: From start of IP through the Study Phase (6 months post-dose) (assessed up to 12 months)
Population: Safety Population. Two participants randomized to placebo group received denosumab by mistake.
Measure: Number; unit: Participants
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 367 | 117
Participants
  Any AEs | 174 | 63
  Any Serious Non-Fatal AEs | 9 | 3
  Any Serious Fatal AEs | 2 | 0

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from start of IP through the Study Phase (6 months post-dose) (assessed up to 12 months).
Description: On-treatment SAEs and non-serious AEs are reported for safety population, comprised of all participants randomized to treatment who received at least one dose of IP.
Groups:
- Denosumab 60mg: Participants received single subcutaneous (SC) injection of denosumab 60 milligrams (mg) at Baseline and Month 6 during the Double-blind Treatment Phase. Particpants also received daily oral supplementation of elemental calcium (at least 600 mg) and vitamin D (at least 400 international unit [IU]).
Arm/Group | Denosumab 60mg | Placebo
Serious Adverse Events (participants affected / at risk) | 11/367 | 3/117
Other Adverse Events (participants affected / at risk) | 43/367 | 24/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab 60mg (N=367) | Placebo (N=117)
Any event (Injury, poisoning and procedural complications) | 3 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Any event (Cardiac disorders) | 1 | 2
Angina unstable (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Any event (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Any event (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Any event (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0
Any event (Nervous system disorders) | 1 | 0
Brain stem infarction (Nervous system disorders) | 1 | 0
Any event (General disorders) | 1 | 0
Sudden cardiac death (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab 60mg (N=367) | Placebo (N=117)
Arthralgia (Investigations) | 24 | 9
Blood cholesterol increased (Investigations) | 19 | 11
Bone density decreased (Investigations) | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.